CLINICAL TRIAL: NCT02627105
Title: The Beef WISE Study: Beef's Role in Weight Improvement, Satisfaction, and Energy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cattlemen's Beef Association, a contractor to the Beef Checkoff (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-0989
Record Dates: First submitted 2015-12-03; First posted 2015-12-10 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Weight Loss
Keywords: weight loss; red meats; obesity; lean body mass; body composition; dietary protein
MeSH Terms: conditions — Weight Loss; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beef group (Experimental): Subjects in this group are asked to consume 4 or more servings of beef per week and to exclude all other red meats from their diet for the 6 month study.
  Interventions: Behavioral: Beef group
- Non-beef group (Other): Subjects in this group are asked to avoid all red meats from their diet for the 6 month study.
  Interventions: Behavioral: Non-beef group

INTERVENTIONS:
Behavioral: Beef group — Subjects in the beef group will be asked to consume 4 or more servings of beef per week (and to avoid all other red meats) during the 6 month study.
  Arms: Beef group
Behavioral: Non-beef group — Subjects in the non-beef group will be asked to avoid all red meats during the 6 month study.
  Arms: Non-beef group

SUMMARY:
This is a 6 month long study to evaluate the inclusion or exclusion of beef within a weight loss program.

DETAILED DESCRIPTION:
This study will compare two protein sources: proteins to include beef as the sole source of red meat compared to proteins excluding red meat within the context of an effective higher-protein weight loss and maintenance program derived from the Colorado Diet.

All subjects will participate in a group-based program consisting of 16 weekly classes in 3-phases designed to produce weight loss and teach participants how to achieve a lifestyle to keep weight off permanently. All groups will be closed (same subjects, same leader) and will consist of 20 participants. Participants in both groups will receive instruction in cooking, recipes, and shopping instruction (using our grocery laboratory). This training will include strategies, tips and preparation techniques for preparing high protein meals according to their assigned groups. All subjects are given exercise plans and all subjects will receive memberships to the Anschutz Health and Wellness Center fitness center for the duration of the study.

After completion of the 16-week program, subjects will be asked to follow the program on their own for an additional 2 months.

This is a randomized study involving 120 study subjects (60 per arm). The investigators will compare the efficacy of inducing weight loss of two treatment arms derived from the Colorado Diet. Subjects will be randomly assigned to one of two study arms and instructed to follow the higher-protein diet by participating in weekly group classes for the first four months of the study. There will be 6 classes of 20 subjects each (three classes for each treatment group). Subjects will be followed in the study for 6 months. Subjects will be randomized into one of two treatment groups as follows:

* Group 1(SOS+B): Subjects will participate in a State of Slim group class, receive a State of Slim book (describing the Colorado Diet), and will receive stipends to be used to help purchase protein food items allowed in the Colorado Diet as modified. The Colorado diet is a high protein (estimated 120-160g/day), low carb and low fat diet. Subjects will be directed and instructed to include beef as their sole source of red meat as a protein source during the study. Subjects will follow the diet protein guidelines, but will be directed and instructed to consume 4 or more servings of beef per week and instructed not to consume any other red meats. Other red meats to be avoided include pork, veal, lamb, buffalo and venison. Subjects will be advised to use the monetary stipends to purchase items from the lists of acceptable foods from the SOS book (to include beef products). Processed beef items will be allowed as identified by a list provided to the subjects.
* Group 2 (SOS): Subjects will participate in a State of Slim class, receive the State of Slim book (describing the Colorado Diet), and will receive stipends to be used to help purchase protein food items allowed in the Colorado diet as modified. Subjects will be directed and instructed to exclude beef and instructed not to consume any other red meats. Other red meats to be avoided include pork, veal, lamb, buffalo, and venison.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 18 - 50 years old
2. BMI of 27 or greater
3. Weight stable (have not lost or gained more than 10 pounds in the last 3 months)
4. Generally healthy
5. Able to exercise 70 minutes per day at moderate intensity
6. Willing and able to participate in a weekly group class for the first 16 weeks of the study and willing to participate in 4 study visits over the 6 month study period

Exclusion Criteria:

1. Pregnant or trying to become pregnant.
2. Diagnosis of type 1 or type 2 diabetes
3. Individuals following a vegetarian/vegan only diet
4. Food allergies (to red meats or other common protein sources)
5. Taking medications that could cause weight loss or weight gain (such as steroids, tricyclic antidepressants, chemotherapy, antipsychotics, prescribed or over the counter weight loss agents). Oral contraceptives can be used as long as subject agrees to not change use of these during the study. Vitamins and minerals which do not have a weight effect are allowed as long as use is continued without change during the study.
6. Current Eating disorder (anorexia or bulimia)
7. Current alcohol or drug abuse or dependence (Subjects who have quit smoking in the last 6 months will be excluded. Smokers whose smoking habits have been stable for the last 6 months and which remain stable during the study can be included).
8. Any medical condition for which following a high protein diet and/or 70 minutes of exercise daily would be inadvisable
9. LDL cholesterol levels above 160 mg/dl or triglycerides above 400 mg/dl.
10. Untreated or unstable hypothyroidism. Thyroid medications must be stable for at least 3 months.

    -

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2015-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in % body weight at the end of a 16 week period and at the end of the 6 month period | 16 weeks and 6 months

SECONDARY OUTCOMES:
Change from baseline in % body fat at the end of a 16 week period | 16 weeks
Change from baseline in lipid panel results at end of 16 week period and end of 6 month period | 16 weeks and 6 months
Change from baseline in fasting blood glucose results at end of 16 week period and end of 6 month period. | 16 weeks and 6 months
Change from baseline in hemoglobin A1C results at end of 16 week period and end of 6 month period. | 16 weeks and 6 months
Differences in responses to study questionnaires between the two groups regarding satisfaction with the weight loss program. | 6 months
Differences in responses to study questionnaires between the two groups regarding adherence to the weight loss program. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: James O Hill, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson GH, Moore SE. Dietary proteins in the regulation of food intake and body weight in humans. J Nutr. 2004 Apr;134(4):974S-9S. doi: 10.1093/jn/134.4.974S. PMID 15051857
- [Background] Anderson GH, Tecimer SN, Shah D, Zafar TA. Protein source, quantity, and time of consumption determine the effect of proteins on short-term food intake in young men. J Nutr. 2004 Nov;134(11):3011-5. doi: 10.1093/jn/134.11.3011. PMID 15514267
- [Background] Barkeling B, Rossner S, Bjorvell H. Effects of a high-protein meal (meat) and a high-carbohydrate meal (vegetarian) on satiety measured by automated computerized monitoring of subsequent food intake, motivation to eat and food preferences. Int J Obes. 1990 Sep;14(9):743-51. PMID 2228407
- [Background] Booth DA, Chase A, Campbell AT. Relative effectiveness of protein in the late stages of appetite suppression in man. Physiol Behav. 1970 Nov;5(11):1299-302. doi: 10.1016/0031-9384(70)90044-2. No abstract available. PMID 5524514
- [Background] Bowen J, Noakes M, Clifton PM. Appetite regulatory hormone responses to various dietary proteins differ by body mass index status despite similar reductions in ad libitum energy intake. J Clin Endocrinol Metab. 2006 Aug;91(8):2913-9. doi: 10.1210/jc.2006-0609. Epub 2006 May 30. PMID 16735482
- [Background] Foster GD, Wyatt HR, Hill JO, McGuckin BG, Brill C, Mohammed BS, Szapary PO, Rader DJ, Edman JS, Klein S. A randomized trial of a low-carbohydrate diet for obesity. N Engl J Med. 2003 May 22;348(21):2082-90. doi: 10.1056/NEJMoa022207. PMID 12761365
- [Background] Latner JD, Schwartz M. The effects of a high-carbohydrate, high-protein or balanced lunch upon later food intake and hunger ratings. Appetite. 1999 Aug;33(1):119-28. doi: 10.1006/appe.1999.0237. PMID 10447984
- [Background] Donnelly JE, Hill JO, Jacobsen DJ, Potteiger J, Sullivan DK, Johnson SL, Heelan K, Hise M, Fennessey PV, Sonko B, Sharp T, Jakicic JM, Blair SN, Tran ZV, Mayo M, Gibson C, Washburn RA. Effects of a 16-month randomized controlled exercise trial on body weight and composition in young, overweight men and women: the Midwest Exercise Trial. Arch Intern Med. 2003 Jun 9;163(11):1343-50. doi: 10.1001/archinte.163.11.1343. PMID 12796071
- [Background] Hill, J. H. & Blundell, J. E. (1986) Macronutrients and satiety: The effects of a high-protein or high-carbohydrate meal on subjective motivation to eat and food preferences. Nutr. Behav. 3: 133-144.
- [Background] Marmonier C, Chapelot D, Louis-Sylvestre J. Effects of macronutrient content and energy density of snacks consumed in a satiety state on the onset of the next meal. Appetite. 2000 Apr;34(2):161-8. doi: 10.1006/appe.1999.0302. PMID 10744905
- [Background] Paddon-Jones D, Westman E, Mattes RD, Wolfe RR, Astrup A, Westerterp-Plantenga M. Protein, weight management, and satiety. Am J Clin Nutr. 2008 May;87(5):1558S-1561S. doi: 10.1093/ajcn/87.5.1558S. PMID 18469287
- [Background] Peters, J.C. Control of Energy Balance. In: Biochemical, physiological, molecular aspects of human nutrition. Second edition, M.H. Stipanuk ed. Saunders Elsevier, 2006, pp. 618-639.
- [Background] Porrini M, Santangelo A, Crovetti R, Riso P, Testolin G, Blundell JE. Weight, protein, fat, and timing of preloads affect food intake. Physiol Behav. 1997 Sep;62(3):563-70. doi: 10.1016/s0031-9384(97)00162-5. PMID 9272665
- [Background] Rolls BJ, Hetherington M, Burley VJ. The specificity of satiety: the influence of foods of different macronutrient content on the development of satiety. Physiol Behav. 1988;43(2):145-53. doi: 10.1016/0031-9384(88)90230-2. PMID 3212049
- [Background] Veldhorst MA, Nieuwenhuizen AG, Hochstenbach-Waelen A, van Vught AJ, Westerterp KR, Engelen MP, Brummer RJ, Deutz NE, Westerterp-Plantenga MS. Dose-dependent satiating effect of whey relative to casein or soy. Physiol Behav. 2009 Mar 23;96(4-5):675-82. doi: 10.1016/j.physbeh.2009.01.004. PMID 19385022
- [Background] Wadden TA, Foreyt JP, Foster GD, Hill JO, Klein S, O'Neil PM, Perri MG, Pi-Sunyer FX, Rock CL, Erickson JS, Maier HN, Kim DD, Dunayevich E. Weight loss with naltrexone SR/bupropion SR combination therapy as an adjunct to behavior modification: the COR-BMOD trial. Obesity (Silver Spring). 2011 Jan;19(1):110-20. doi: 10.1038/oby.2010.147. Epub 2010 Jun 17. PMID 20559296
- [Background] Westerterp-Plantenga MS, Nieuwenhuizen A, Tome D, Soenen S, Westerterp KR. Dietary protein, weight loss, and weight maintenance. Annu Rev Nutr. 2009;29:21-41. doi: 10.1146/annurev-nutr-080508-141056. PMID 19400750
- [Result] Sayer RD, Speaker KJ, Pan Z, Peters JC, Wyatt HR, Hill JO. Equivalent reductions in body weight during the Beef WISE Study: beef's role in weight improvement, satisfaction and energy. Obes Sci Pract. 2017 Jul 11;3(3):298-310. doi: 10.1002/osp4.118. eCollection 2017 Sep. PMID 29071106
- [Result] Sayer RD, Peters JC, Pan Z, Wyatt HR, Hill JO. Hunger, Food Cravings, and Diet Satisfaction are Related to Changes in Body Weight During a 6-Month Behavioral Weight Loss Intervention: The Beef WISE Study. Nutrients. 2018 May 31;10(6):700. doi: 10.3390/nu10060700. PMID 29857497
- [Derived] Clina JG, Pan Z, Wyatt HR, Peters JC, Hill JO, Sayer RD. Secondary analysis of a university-based weight loss program in on-campus versus off-campus employees. Obes Sci Pract. 2022 Jun 4;8(6):767-774. doi: 10.1002/osp4.618. eCollection 2022 Dec. PMID 36483127